CLINICAL TRIAL: NCT06047223
Title: Analysis of Brain Diffusion Tensor Image in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle investigator, Bundang CHA Hospital
Other Study IDs: 2023-08-005
Record Dates: First submitted 2023-08-28; First posted 2023-09-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic resonanace imaging — Magnetic resonance imaging for measurement of diffustion tensor imaging

SUMMARY:
This clinical study aims to confirm the characteristics of the functional ansiotropy value according to the individual characteristics of stroke patients by taking brain diffusion tensor images for stroke patients and using the MRI. To compare hematologic indicators and neurological function levels of stroke patients at the time of imaging examination with brain diffusion tensor imaging indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20 years or older with a history of stroke
2. After hearing a detailed explanation of this study and fully understanding it, the subject or legal representative voluntarily decides to participate and agrees in writing to observe the precautions

Exclusion Criteria:

Patients who meet one or more of the following cannot participate in the study.

1. Those with severe medical conditions such as unstable conditions in the cardiovascular system, digestive system, respiratory system, endocrine system, etc., and those with poor general health
2. In the case of a person with impaired consent, a person without a guardian
3. Patients who have devices that may be affected by MRI, such as pacemakers, spinal cord stimulators, cochlear implants, VP shunts, and nerve stimulators, inserted into the body
4. Other cases where the researcher judges that participation in this study is not suitable (This study is not an interventional study, and patients who are participating in other clinical trials or studies or who have participated in other clinical trials or studies within the past 30 days can also participate in this study.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of magnetic resonanace imaging (MRI) | Through study completion, an average of 1 day
  MRI scan is a process of measuring changes of diffusion tensor tractography

SECONDARY OUTCOMES:
Measurement of Korean version of coma recovery scale-revised (K-CRSR) | Through study completion, an average of 1 day
  K-CRSR is Korean version of standardized neurobehavioral assessment measure designed for use in patients with disorders of consciousness. he scale is intended to be used to establish diagnosis, monitor behavioral recovery, predict outcome, and assess treatment effectiveness.
Measurement of Korean version of Montreal Cognitive Assessment (K-MoCA) | Through study completion, an average of 1 day
  K-MoCA is a measurement to evaluate the memory loss or other symptoms of cognitive decline. It contains 30 questions and taskes around to 12 minutes to complete. Scores range from 0 to 30. A score of 26 and higher is considered normal.
Measurement of clinical dementia rate (CDR) | Through study completion, an average of 1 day
  CDR is a rating scale for staging patients diagnosed with dementia. The CDR evaluates cognitive, behavioral and functional aspects of Alzheimer disease and other dementias. It is calculated on the basis of testing six different cognitive and behavioral domains such as memory, orientation, judgment and problem sloving, community affairs, home and hobbies performance, and personal care. The CDR is based on a scale of 0-3: no dementia (CDR = 0), questionable dementia (CDR = 0.5), MCI (CDR = 1), moderate cognitive impairment (CDR = 2) and severe cognitive impairment (CDR = 3)
Measurement of Korean version of oxford cognitive screen (OCS-K) | visit 1
  OCS is an assessment of major cognitive domains of memory, language, number, praxis, executive functions and attention.
Measurement of digit span test. | Through study completion, an average of 1 day
  Digit span test is a measurment to assess the storage capacity of a person's working memory. A testperson is visually or auditorily to a sequence of digits on after another. Right afterwards, the test subject has to recall the correct digits in the same order.
Measurement of digit span test. | Through study completion, an average of 1 day
  inhibit cognitie interference. The stroop test consists of colors that are writen in words but in the wrong color ink, The test-taker has to be able to state the color that the word is written in and be able to ignore whatever the actual word is.
Measurement of Korean version of western aphasia battery (K-WAB) | Through study completion, an average of 1 day
  K-WAB is designed as an assessment tool to examine linguistic skills (information content, fluency, auditory comprehension, repetition, naming and word finding, reading, and writing) and main nonlinguistic skills (drawing, block design, calculation, and praxis) of adults with aphasia.
Measurement of motricity index (MI) | Through study completion, an average of 1 day
  MI is a process of the evaluating the function and strength of upper, lower extremities and trunk in score.
Measurement of berg balance scale (BBS) | Through study completion, an average of 1 day
  BBS is a measurement of balancing function. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total score = 56
Measurement of functional ambulatory category (FAC) | Through study completion, an average of 1 day
  FAC is a measurement of a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use personal assistive device.
Measurement of time up and go (TUG) | Through study completion, an average of 1 day
  TUG is a measurement of a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. 11-20 seconds are within normal limits for frail elderly and disables patients, and greater than 20 seconds means the person needs assistance outside and indicates further examintaiton and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
Measurement of Fugl-Meyer assessment (FMA) | Through study completion, an average of 1 day
  FMA is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sesation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research determine disease severity, describe motor recovery, and to plan and assess treatment.
Measurement of action research arm test (ARAT) | Through study completion, an average of 1 day
  ARAT is a 19 item observational measurement to assess upper extremity performance (coordination, dexterity and functioning). Items comprising ARAT are categorized into four subscales (grasp, grip, pinch and gross movement). Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performend normally)
Measurement of Korean version of modified barthel index (K-MBI) | Through study completion, an average of 1 day
  MBI is a measurement of degree of independence of a patient from any assistance. It covers 10 domains of daily activities: bowel and bladder control, grooming, toilet use, feeding, trasnfers, walking, dressing, climbing stairs and bathing
Measurement of motion analysis | Through study completion, an average of 1 day
  Motion analysis is a process of measuring and evaluating gait function in kinetic parameters of range of motion in angle of each joint by degree throguh Qualisys motion analysis system
Measurement of motion analysis | Through study completion, an average of 1 day
  Motion analysis is a process of measuring and evaluating gait function and kinematic parameters including moment (Nm/kg) of each joint throguh Qualisys motion analysis system
Measurement of motion analysis | Through study completion, an average of 1 day
  Motion analysis is a process of measuring and evaluating gait function and kinematic parameters including power (Nm/s*kg) of each joint throguh Qualisys motion analysis system
Measurement of motion analysis | Through study completion, an average of 1 day
  Motion analysis is a process of measuring and evaluating gait function and kinematic parameters including ground reaction force (N/kg) of each joint throguh Qualisys motion analysis system

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — Bundang CHA Hospital
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea